CLINICAL TRIAL: NCT03652974
Title: Disturbance of Plasma Cytokine Parameters in Clozapine-Resistant Treatment-Refractory Schizophrenia (CTRS) and Their Association With Combination Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Pudong New Area Mental Health Center (Unknown); The Affiliated Brain Hospital of Guangzhou Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 81171272
Record Dates: First submitted 2018-08-25; First posted 2018-08-31 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia， clozapine， amisulpride, valproate， ECT, cytokine
MeSH Terms: conditions — Schizophrenia | interventions — Valproic Acid; Clozapine; Amisulpride

STUDY DESIGN:
Intervention Model Description: Drug: amisulpride, sodium valproate , placebo and Clozapine amisulpride, sodium valproate and placebo may be used as a synergistic agent of clozapine in the treatment of treatment-resistant schizophrenia Other Name: Valproate Device: modified electroconvulsive therapy(MECT) with Clozapine modified electroconvulsive therapy(MECT) may be used as a synergistic agent of clozapine in the treatment of treatment-resistant schizophrenia Device: Modified electroconvulsive therapy(MECT) with Clozapine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sodium valproate with clozapine (Experimental): sodium valproate, dosage form: 250 mg, dosage and frequency:250 mg/d for 1 week, 500 mg/d for week 2 , 1000 mg/d for weeks 3, 4, 5, 6, 7 , 8, 9, 10, 11and 12; clozapine, dosage and frequency:300~600 mg/d; duration: 12 weeks.
  Intervention: Drug: sodium valproate with Clozapine
  Interventions: Drug: sodium valproate with Clozapine
- Modified electroconvulsive therapy with clozapine (Experimental): 12 times MECT for 12 weeks，once a week for the 12 weeks; clozapine, dosage and frequency:300~600 mg/d; duration: 12 weeks.
  Intervention: Device: modified electroconvulsive therapy(MECT) with Clozapine
  Interventions: Device: modified electroconvulsive therapy(MECT) with Clozapine
- amisulpride (Experimental): amisulpride, dosage form: 200 mg, dosage and frequency:200 mg/d for 1 week, 400 mg/d for week 2,800 mg/d for weeks 3, 4, 5, 6, 7 , 8, 9, 10, 11and 12; clozapine, dosage and frequency:300~600 mg/d; duration: 12 weeks.
  Intervention: Drug: amisulpride with Clozapine
  Interventions: Drug: amisulpride with Clozapine
- placebo (Placebo Comparator): The amisulpride and placebo tablets were identical in appearance. One placebo tablet for the first one week, two placebo tablets for the second week, four placebo tablets for weeks 3, 4, 5, 6, 7 , 8, 9, 10, 11and 12; clozapine, dosage and frequency:300~600 mg/d; duration: 12 weeks.
  Intervention: Drug: placebo with Clozapine
  Interventions: Drug: placebo with Clozapine

INTERVENTIONS:
Drug: sodium valproate with Clozapine — sodium valproate may be used as a synergistic agent of clozapine in the treatment of treatment-refractory schizophrenia
  Other Names: Valproate
  Arms: sodium valproate with clozapine
Device: modified electroconvulsive therapy(MECT) with Clozapine — modified electroconvulsive therapy(MECT) may be used as a synergistic agent of clozapine in the treatment of treatment-refractory schizophrenia
  Arms: Modified electroconvulsive therapy with clozapine
Drug: amisulpride with Clozapine — amisulpride may be used as a synergistic agent of clozapine in the treatment of treatment-refractory schizophrenia
  Arms: amisulpride
Drug: placebo with Clozapine — placebo may be used as a synergistic agent of clozapine in the treatment of treatment-refractory schizophrenia
  Arms: placebo

SUMMARY:
In this study, investigators designed a double-blind randomized trial to compare the efficacy and safety between sodium valproate, amisulpride and MECT combination therapy in clozapine-treated refractory schizophrenia (CTRS).

DETAILED DESCRIPTION:
Schizophrenia is one of the most serious mental illnesses worldwide that affects approximately 1% of the worldwide population and result in a heavy economic burden to affected family. Antipsychotics are the main stay of treatment of schizophrenia, however, there are still approximately 1/3 schizophrenia patients who does not responded to the antipsychotic agents, and these patients easily develop into treatment-refractory schizophrenia (TRS).

Clozapine is the only evidence based effective medication for treatment-refractory schizophrenia (TRS). In spite of its prominent efficacy, approximately 1/3-2/1 treatment-refractory schizophrenia (TRS) treated with clozapine still present with significant residual psychotic symptoms and negative symptoms. As such, over time, clinicians struggled to find strategies to improve outcome by augmenting the concomitant psychiatric treatments, including not only combining antipsychotics but also combining a mood stabilizer or electroconvulsive therapy (ECT).

Clozapine is an antipsychotic drug with multi receptor blocking effect and has a low affinity for dopamine D2. Studies of traditional antipsychotics have suggested that maximal efficacy occurs with dopamine D2 occupancy of 70% or more, while clozapine's dopamine D2 occupancy levels less than 60%. Amisulpride has a highly selective blocking effect on dopamine D2 and dopamine D3 receptors and has no affinity for any other known receptors. Its unique dopamine receptor blocking effect may selectively enhances the limited dopamine D2 blocking effect of clozapine, making it possible to be a suitable and effective drug for combination with clozapine. A number of promising studies that have augmented clozapine with amisulpride, have shown psychiatric symptoms improvement in TRS versus those on clozapine alone.

Both electroconvulsive therapy (ECT) and antiepileptic drugs, such as sodium valproate, shares anticonvulsant properties and anticonvulsant effect relate to clinical efficacy. In 1983, Sackeim et al. pointed out that electroconvulsive therapy (ECT)-induced cortical gamma-aminobutyric-acid (GABA) depletion may be the reason for its anticonvulsant action. In addition, the effect of electroconvulsive therapy (ECT) on the gamma-aminobutyric-acid (GABA) system was confirmed by several studies. Interestingly, it has been reported that the therapeutic effect of sodium valproate combined with antipsychotics is closely related to gamma-aminobutyric-acid (GABA) system.

Growing evidence suggests that the immune, endocrine, and nervous systems interact with each other through cytokines, hormones, and neurotransmitters. The activation of the immune system may be involved in the neuropathological changes occurring in the central nervous system. Among several components of immune pathogenesis, aberrant cytokine signaling is considered as one of the key contributors. Many cytokines have been speculated to be involved in the pathological process of schizophrenia. IL-2 acts as a growth factor for T cells, NK cells and B cells, abnormalities of IL-2 serum levels or its production were found in acute schizophrenia cases. IL-6 is an inflammatory cytokine, which plays significant role in neurobiological functions like neuronal differentiation and survival, synaptic transmission and brain morphometry. The abnormal expression of IL-6 can be found in both first-episode and chronic schizophrenia. TNF-α is one of the most important pro-inflammatory cytokines, which expressed mainly by macrophages. Previous studies have found that the expression of TNF-α is abnormal in patients with schizophrenia.

The primary objective of this study was to compare the efficacy and safety between sodium valproate, amisulpride and MECT combination therapy in clozapine-treated refractory schizophrenia during a 12 weeks period. In addition, the effect of combined therapy on plasma cytokines (IL-2, IL-6 and TNF-α) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* 18～60 years old
* Clozapine resistance was defined as used at least two antipsychotics with different chemical structures with appropriate dosages for a sufficient duration, and recently have received stable dose of clozapine 400 mg or more per day for at least 6 months.
* Signed an informed consent

Exclusion Criteria:

* Patients to be diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) for substance abused, development delayed
* Suffering from serious physical disease and can not accept the treatment
* Allergic to sodium valproate, amisulpride, propofol, succinylcholine or atropine
* Participated in any clinical subject within 30 days
* Pregnancy or lactation
* Inability to sign informed consent because of capacity due due to severe mental illness, significant psychomotor agitation or slowness test completion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | the baseline
  The battery of Positive and Negative Syndrome Scale (PANSS) test will be administered in a 30-minute sessions to evaluate the psychiatric symptoms.
Positive and Negative Syndrome Scale (PANSS) | the end of the six week
  The battery of Positive and Negative Syndrome Scale (PANSS) test will be administered in a 30-minute sessions to evaluate the psychiatric symptoms.
Positive and Negative Syndrome Scale (PANSS) | the end of the twelve week
  The battery of Positive and Negative Syndrome Scale (PANSS) test will be administered in a 30-minute sessions to evaluate the psychiatric symptoms.
Scale for the Assessment of Negative Symptoms (SANS) | the baseline
  The Scale for the Assessment of Negative Symptoms (SANS) was applied to assess negative symptoms.
Scale for the Assessment of Negative Symptoms (SANS) | the end of the six week
  The Scale for the Assessment of Negative Symptoms (SANS) was applied to assess negative symptoms.
Scale for the Assessment of Negative Symptoms (SANS) | the end of the twelve week
  The Scale for the Assessment of Negative Symptoms (SANS) was applied to assess negative symptoms.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | the baseline
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) was used to evaluate the cognitive performance.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | the end of the six week
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) was used to evaluate the cognitive performance.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | the end of the twelve week
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) was used to evaluate the cognitive performance.
Clinical Global Impression (CGI) | the baseline
  The Clinical Global Impression (CGI) including severity scale (CGI-S), improvement scale (CGI-I), and efficacy index (CGI-E) was used to evaluate the severity of symptoms and treatment response and treatment effect, respectively.
Clinical Global Impression (CGI) | the end of the six week
  The Clinical Global Impression (CGI) including severity scale (CGI-S), improvement scale (CGI-I), and efficacy index (CGI-E) was used to evaluate the severity of symptoms and treatment response and treatment effect, respectively.
Clinical Global Impression (CGI) | the end of the twelve week
  The Clinical Global Impression (CGI) including severity scale (CGI-S), improvement scale (CGI-I), and efficacy index (CGI-E) was used to evaluate the severity of symptoms and treatment response and treatment effect, respectively.
Treatment Emergent Symptom Scale (TESS) | the baseline
  The Treatment Emergent Symptom Scale (TESS) was used to assess the severity of treatment adverse events.
Treatment Emergent Symptom Scale (TESS) | the end of the six week
  The Treatment Emergent Symptom Scale (TESS) was used to assess the severity of treatment adverse events.
Treatment Emergent Symptom Scale (TESS) | the end of the twelve week
  The Treatment Emergent Symptom Scale (TESS) was used to assess the severity of treatment adverse events.
plasma cytokines IL-2, IL-6 and TNF-α | the baseline
  The plasma cytokines IL-2, IL-6 and TNF-α would be measured using ELISA kits (R & D Systems, Mississauga, Ontario, CANADA).
plasma cytokines IL-2, IL-6 and TNF-α | the end of the twelve week
  The plasma cytokines IL-2, IL-6 and TNF-α would be measured using ELISA kits (R & D Systems, Mississauga, Ontario, CANADA).

CONTACTS AND LOCATIONS:
Overall Officials: Zezhi Li, M.D., Principal Investigator — Department of Psychiatry, The Affiliated Brain Hospital of Guangzhou Medical University
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu MH, Liu ZJ, Hu QY, Yang JY, Jin Y, Zhu N, Huang Y, Shi DH, Liu MJ, Tan HY, Zhao L, Lv QY, Yi ZH, Wu FC, Li ZZ. Amisulpride augmentation therapy improves cognitive performance and psychopathology in clozapine-resistant treatment-refractory schizophrenia: a 12-week randomized, double-blind, placebo-controlled trial. Mil Med Res. 2022 Oct 18;9(1):59. doi: 10.1186/s40779-022-00420-0. PMID 36253804